CLINICAL TRIAL: NCT05801211
Title: Colonic Resection, stOma, or Self-expandable Metallic Stent for obstruCtive Left cOlon Cancer. The CROSCO-1 Multicenter, Prospective Cohort Study
Brief Title: Colonic Resection or Stoma, or Self-expandable Metallic Stent for obstruCtive Left cOlon Cancer
Acronym: CROSCO-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Sanitaria di Firenze (Other)
Responsible Party: Principal Investigator, Alessio Giordano, Principal Investigator, Azienda Sanitaria di Firenze
Other Study IDs: Alessio Giordano
Record Dates: First submitted 2023-03-08; First posted 2023-04-06 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Colon Cancer
Keywords: SEMS; obstructive CRC; primary anastomosis; Hartmann
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- primary surgical tumor resection with anastomosis or only tumor resection without anastomosis: primary surgical tumor resection with a primary colorectal anastomosis (associated or not with a diverting loop ileostomy) or without a primary anastomosis ("Hartmann's procedure")
  Interventions: Procedure: primary tumor resection
- endoscopic stent positioning: staged resection after endoscopic stenting with Self-expandable Metallic Stent (SEMS)

INTERVENTIONS:
Procedure: primary tumor resection — primary surgical tumor resection with a primary colorectal anastomosis (associated or not with a diverting loop ileostomy) or without a primary anastomosis ("Hartmann's procedure")
  Groups: primary surgical tumor resection with anastomosis or only tumor resection without anastomosis

SUMMARY:
CROSCO-1 study is a national, multi-center, prospective observational study presenting patients to the emergency departments of the participating centers with obstructive left colon cancer (in the absence of metastases and peritoneal carcinomatosis) undergoing primary surgical tumor resection with a primary colorectal anastomosis (associated or not with a diverting loop ileostomy) or without a primary anastomosis ("Hartmann's procedure") or staged resection after endoscopic stenting with Self-expandable Metallic Stent (SEMS).

The main questions it aims to answer are:

* the Stoma rate at 1 year after tumor resection
* the 30-day and 90-day major morbidity and mortality
* 1-year quality of life (EQ-5D-5L test)
* Timing of chemotherapy initiation and type of chemotherapy regimen. Participants will have an obstructive left colon cancer localized (no peritoneal carcinosis or distant metastasis).

Researchers will compare: primary surgical tumor resection with a primary colorectal anastomosis (associated or not with a diverting loop ileostomy) or an "Hartmann's procedure" with a staged resection after endoscopic stenting with SEMS.

DETAILED DESCRIPTION:
Since surgical and oncological outcomes of the different treatment strategies for obstructing left colon cancers have not been studied on a large scale globally, we launched the CROSCO-1 study intending to compare the clinical results of all these therapeutic regimens in a cohort of patients treated for obstructive left-sided colorectal cancer (CRC).

The primary aim of the CROSCO-1 (Colonic Resection, stOma or self-expanding metal Stents for obstruCtive left cOlon cancer) study is to describe the outcomes of the management of emergency presentations of obstructive left CRC with colorectal resection with or without primary anastomosis versus the staged approach with SEMS insertion and subsequent colorectal resection. The primary aim of the CROSCO-1 study will be the 1-year stoma rate of patients undergoing primary emergency surgical resection (Hartmann procedure or primary resection and anastomosis) compared with patients undergoing staged resection (emergency endoscopic treatment with SEMS followed by elective resection). Other outcomes will be 30-day and 90-day major morbidity and mortality, 1-year quality of life, and the timing and type of chemotherapy initiation in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, ≥ 18 years old.
2. Patients with abdominal CT scan diagnosis of colonic obstruction due to obstructive left colonic cancer (sigmoid or descending colon).
3. Absence of distant metastases on abdominal and chest CT scan.
4. Patients who may face a one-year follow-up.
5. Patients fit for surgery.
6. Patients with colonic adenocarcinoma on postoperative histological examination.

Exclusion Criteria:

1. Right-side or trasverse colon cancer.
2. Surgical or endoscopic palliation in patients with peritoneal carcinomatosis, locally advanced Colorectal cancer (CRC) (T4 sec. TNM), M1 disease.
3. Bowel obstruction determinated by other tumors or benign inflammatory stenosis.
4. Concomitant bowel abscess, perforation, or fistula.
5. Elective procedures.
6. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all consecutive adult patients (≥18 years of age) presenting acutely ( unplanned and non-elective presentation to hospital for urgent or emergency reasons) at the participating centers with a clinical and radiological diagnosis of (known or unknown descending or sigmoid colon tumor) for 1 year. According to the different management methods, the cohort will be divided into the following categories:
  1. Primary tumor resection, which will include patients treated with Hartmann's procedure or primary resection with anastomosis (with or without a diverting ileostomy).
  2. Staged tumor resection, which will include patients treated with a Self-expandable Metallic Stent (SEMS) insertion, followed by colorectal resection.
Sampling Method: Non-Probability Sample
Enrollment: 434 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Stoma rate at 1 year after tumor resection | 1 year
  the number of stomas after 1 year of primary surgery with tumor resection

SECONDARY OUTCOMES:
30-day and 90-day major morbidity | 30-days; 90-days
  morbidity after 30 and 90-days
30-day and 90-day mortality | 30-days; 90-days
  mortality (Overall survival) after 30 and 90-days
1-year quality of life (The 5-level EQ-5D version (EQ-5D-5L)test) | 1-year
  The EQ-5D-5L is an instrument to describe the quality of life with a state system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. In this first part, the patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions with graduate answers from 1 (no problem) to 5 (extreme limitations). The aggregation of the responses forms a five-digit number representing the patient's health status. in the second part, the patient is asked to indicate an assessment using a visual analog (VAS) graphically represented by a graduated scale ranging from 0 (the worst possible state of health) to 100 (the best possible state of health) on which the interviewee indicates his or her perceived level of health.
Timing of chemotherapy initiation | 2-years
  data for chemotherapy initiation in both groups of study
type of chemotherapy regimen | 2-years
  type of drugs regimen in both groups of study

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Giordano, Principal Investigator — AOU Careggi Firenze

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD can be Share for 1 year after follow up closure
Access Criteria: by email with colleagues who will be interested